CLINICAL TRIAL: NCT02031588
Title: Impact of Ceftriaxone and/or Fluoroquinolone (FQ) Treatment on the Gut Microbiota of Hospitalized Patients.
Acronym: EVOTAR
Status: Terminated | Type: Observational
Why Stopped: lack of recruitement
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: RAFREU53
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Bacterial Infections
Keywords: Study of commensal flora; Fluoroquinolones
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples will be collected on 4 separate days for patients treated with antibiotics:
  T0: before treatment begins T1: at the end of treatment or discharge from the hospital T2: 3-6 months after the end of treatment T3: 10-14 months after the end of treatment For patients receiving sequentially ceftriaxone followed by a FQ, an additional sample will be collected at the end of ceftriaxone treatment.
  In the reference group, stool samples will be collected:
  T0: at inclusion in the study T1: at hospital discharge The purpose is to study the bacterial DNA contained in the stool. No analysis will be performed on the human patient DNA.
  Changes in the gut microflora will be analysed by metagenomics deep sequencing performed by Dushko Ehrlich (INRA, France).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Ceftriaxone: Patients receiving a C3G (ceftriaxone) during the hospitalization.
- Ceftriaxone + Fluoroquinolone: ceftriaxone followed by fluoroquinolone (which is a common situation in clinical practice, Fluoroquinolone being prescribed after obtaining antibiogram).
- Fluoroquinolones: fluoroquinolones (levofloxacin, ofloxacin, moxifloxacin or ciprofloxacin).
- Reference: A third reference group will consist of patients hospitalized in the same services as the "case" patients but did not receive antibiotics (60 patients). They will have an idea of possible changes in flora during hospitalization without any antibiotics, for example due to horizontal transfer of resistant strains. This group will be composed of 60 patients who had not received antibiotics within 3 months before and not receiving for the duration of their participation.

SUMMARY:
Observational study of the effects of antibiotics on commensal flora. Realization of stool samples and nasal swabs before and after antibiotic therapy.

DETAILED DESCRIPTION:
The emergence of resistance to fluoroquinolone (FQ) and is a major problem worldwide. The commensal flora is the main reservoir for antibiotic resistance. Understanding the factors (environmental, patient-related, dosis-related, drug-related…) involved in the emergence of resistance to fluoroquinolones in the commensal flora of patients treated with a FQ, may help prevent it and preserve the efficiency of these important antibiotics. Samples of digestive flora will be collected from hospitalized patients before receiving a FQ or Ceftriaxone, at the end of the treatment and 3 month after the end of treatment. Clinical data will be collected.

ELIGIBILITY:
Inclusion criteria for the patients treated with antibiotics

* Adult patient hospitalized in a participating ward of the hospital for an expected duration of more than 24 hours.
* Treatment by ceftriaxone and / or a fluoroquinolone started by the attending physicians during hospitalization.
* No hospitalization or stay in nursing home in the previous three months.
* No use of antibiotics in the last 3 months
* Not receiving other antibiotics than ceftriaxone or FQ
* Informed consent

Inclusion criteria for the patients in the reference group

* Adult patient hospitalized in a participating ward of the hospital for an expected duration of more than 24 hours.
* Not receiving any antibiotic and not expected to receive any during hospitalization
* No hospitalization or stay in nursing home in the previous three months.
* No use of antibiotics in the last 3 months
* Informed consent

Exclusion criteria

* Pregnant or nursing women
* Patient who underwent colectomy or suffering from chronic intestinal disease (inflammatory intestinal disease or short bowel syndrome)
* Patient who used a bowel preparation solution for colonoscopy during hospitalization or in the previous week.
* Protected adult patient (deputyship or guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Hospitalized patients treated with ceftriaxone and / or an oral fluoroquinolone at Beaujon hospital, Clichy, France.
  * A reference group of hospitalized patients not receiving antibiotics, hospitalized in the same wards as the treated patients
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Describe the changes in the composition of the gut microbial flora in relation to the initial flora (T0) in patients receiving antibiotics, by date of sampling, treatment received, dose, duration of therapy, ward, and duration of hospital stay. | 1 year
  The primary endpoint is the change in composition of the microbial flora in relation to the initial flora (T0), at the exit of the hospital or at the end of treatment if occurs while the patient is still hospitalized (bis T0, T1, T1 bis), 3 months after the end of treatment (T2) and one year after the end of treatment (T3).

SECONDARY OUTCOMES:
A secondary endpoint is to describe the changes in the gut microbiota of hospitalized patients not receiving antibiotics. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Victoire De Latours, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France